CLINICAL TRIAL: NCT07212530
Title: "Promoting Health in Adolescents With and Without Chronic Diseases Through Emotional Development: Design and Implementation of a Serious Game Technology Platform (EmoTIChealth)"
Brief Title: EmoTIChealth: Promoting Adolescent Health Through a Serious Game.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Universitat Politècnica de València (Other)
Responsible Party: Principal Investigator, M. Antonia Pérez-Marín, Associate Professor, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EmoTIChealth
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes; Asthma; Allergic Rhinitis; Food Allergy; Adolescent Development
Keywords: Type 1 Diabetes; Asthma; Allergic Rhinitis; Food allergy; Serious Game; Technology platform; Psychological intervention; Adolescence; Quality of life; chronic organic illnesses; Socioemotional Education; Health Promotion
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Asthma; Rhinitis, Allergic; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Adolescents who receive the treatment program will previously constitute their own control group (waiting list control group). Thus, diagnostic measures will be obtained in all of them in an initial evaluation (T1), and after 4 weeks of this assessment the treatment program will be started. In the first contact session, 4 weeks after T1, all adolescents will be reassessed (T2), and after this, the treatment program will be started (within an estimated time of 10 days maximum from this second pre-treatment evaluation, the estimated duration of play/treatment being 4 weeks). After the completion of the serious game, a new asssesment pass will be performed (T3) in order to review the post-treatment change. Thus, the estimated time between T2 and T3 will be equivalent to that between T1 and T2, being 4 weeks.
  Interventions: Behavioral: EmoTIChealth

INTERVENTIONS:
Behavioral: EmoTIChealth — The EmoTIChealth technological platform intervenes in users through a "serious game", i.e. a video game whose main purpose is to teach or provide the player with certain skills that serve to achieve a higher purpose than the game itself. The game is composed of 6 areas, each of which refers to one of the variables that are analyzed or considered important in promoting health related quality of life and adaptation to chronic illness: Area 1. Psychoeducation; 2. Emotional awareness and expression; 3. Emotional regulation; 4. Problem solving; 5. Self-esteem and identity;6. Social skills and communication.

SUMMARY:
The intervention program targets adolescents between 12 and 16 years of age. The intervention program is designed for adolescents during a critical developmental stage marked by significant life transitions, where building strong personal resources and receiving psychological support is essential to foster socioemotional skills and overall well-being. The serious game aims to promote psycho-emotional health in the general adolescent population, supporting healthy development and preventing future emotional difficulties. At the same time, it incorporates specific modules for adolescents living with chronic conditions such as asthma, food allergy, type 1 diabetes, and allergic rhinitis, who may face additional risks of psychological challenges that can complicate treatment and prognosis. By combining universal health promotion with tailored support, the program addresses both the needs of healthy adolescents and those with chronic illnesses.

The platform integrates digital and technological tools for dynamic and personalized intervention. Artificial intelligence adapts activities and feedback to each participant's socio-demographic profile and evolving needs, this supports directly in participants' daily lives and natural environments, making the experience more relevant and impactful. The serious game, proven effective in engaging young people, goes beyond traditional psychoeducation by creating an interactive environment where adolescents develop socio-emotional competencies, resilience, and health-related knowledge. Through its six thematic areas, the game promotes overall well-being and healthy habits, while its condition-specific modules provide targeted guidance and coping strategies for asthma, food allergies, type 1 diabetes, and allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by parents/guardians and participants.
* Aged between 12 and 16 years old

Exclusion Criteria:

* No access to internet or new technologies
* Not a Spanish speaker.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Change Quality of Life (Baseline-Pre-Post) | Baseline up to 8 weeks
  KIDSCREEN-27. This scale consists of 27 items in 5 subscales. Physical well-being, mood, family life, school life, peer relations. Scores range from 27 to 135. Higher scores indicate a higher quality of life in general and in each of the subscales.
  First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 4 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 4 weeks after the second measurement, the third measurement of the same variable was carried out. [Time Frame: Baseline up to 8 weeks]
Change Emotional and Behavioral Problems (Baseline-Pre-Post) | Baseline up to 8 weeks
  SDQ: This questionnaire is used to assess the possible presence of psychopathology and the emotional and behavioral adjustment of adolescents. It is a 25-item Likert-type (1-3) questionnaire. The items of this questionnaire are divided into 5 subscales: emotional symptomatology, conduct problems, hyperactivity, peer problems and prosocial behavior. Higher scores on each scale indicate greater difficulties.
  First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 4 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 4 weeks after the second measurement, the third measurement of the same variable was carried out.
Change Emotional Competences (Baseline-Pre-Post) | Baseline up to 8 weeks
  EAQ-30: This questionnaire consists of 30 Likert-style items (1-False to 3-True), and aims to identify how adolescents think about their feelings, as well as the degree to which they feel them and the ability to express them. In addition to an overall score, this tool is composed of 6 subscales that attempt to describe different aspects of emotional functioning. Higher scores indicate greater use of emotional awareness and regulation strategies.
  First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 4 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 4 weeks after the second measurement, the third measurement of the same variable was carried out.
Change Self-concept (Baseline-Pre-Post) | Baseline up to 8 weeks
  CAG: This questionnaire aims to measure self-concept in adolescents from a multidimensional perspective. It consists of 48 Likert-type response items ranging from 1 to 5, providing a score range of 48 to 240. Physical Self-Concept, Social Acceptance, Family Self-Concept, Intellectual Self-Concept, Personal Self-Assessment, and Sense of Control. The questionnaire provides an overall self-concept score, as well as scores for 6 subdimensions: Higher scores indicate higher self-concept.
  This is the first measurement. After obtaining the participant's informed consent, we assessed the initial score for this outcome.
  The second measurement, labeled PRE, was conducted up to 4 weeks after the first measurement of the same variable.
  The third measurement, labeled POST, was carried out up to 4 weeks after the second measurement.
Change Coping (Baseline-Pre-Post) | Baseline up to 8 weeks
  Social Problem-Solving Inventory- Revised (SPSI-R). This questionnaire attempts to reflect the cognitive, affective and behavioral responses to the problems of daily life or the different difficulties we try to solve. This reduced version consists of 25 Likert-type items, grouped into the following 5 dimensions: Rational problem solving, Avoidant style, Impulsive style, Positive problem orientation and Negative problem orientation. Higher scores on each dimension signify the coping style used by the adolescent.
  First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 4 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 4 weeks after the second measurement, the third measurement of the same variable was carried out.
Change Social Skills (Baseline-Pre-Post) | Baseline up to 8 weeks
  CHASO: It consists of 40 Likert-type response items ranging from 1 to 5 (1 - Very uncharacteristic of me; 5 - Very characteristic of me) and assesses a total of 10 skills: 1. Interacting with strangers; 2. Dealing with criticism; 4. Interacting with people I am attracted to; 5. Staying calm in the face of criticism; 6. Public speaking/interacting with superiors; 7. The scores for each of these skills are calculated from the sum of the items that make them up. Higher scores indicate higher social skills.
  First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 4 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 4 weeks after the second measurement, the third measurement of the same variablewas carried out.

SECONDARY OUTCOMES:
Change in Perception of Threat of disease(Baseline-Pre-Post) | Baseline up to 8 weeks
  The Brief Illness Threat Questionnaire (BIP-Q) is used, which consists of 5 items with a Likert scale from 0 to 10. This questionnaire mainly assesses consequences of the illness, duration of the illness, identity, worry about the illness and emotional impact of the illness. The scale is interpreted so that the higher the score, the greater the sense of perceived threat.
  First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 4 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 weeks after the second measurement, the third measurement of the same variable was carried out.
Change Psychoeducation Diabetes | Start of the intervetion and during it.
  Psychoeducation of the disease: the ECODI Diabetes knowledge scale will be used to assess this variable. This scale consists of 25 items and four dimensions: basic knowledge and self-care, laboratory values, diet and physical exercise. It is a scale that is corrected by the number of hits and misses. Psychoeducation about the disease: The ECODI diabetes knowledge scale is used to assess this variable. This scale consists of 25 items and four dimensions: basic knowledge and self-care, laboratory values, diet and exercise. It is a scale that is corrected by the number of hits and misses.
Change Resilience (Baseline-Pre-Post) | Baseline up to 8 weeks
  Connor-Davidson Resilience Scale to assess the ability to cope with stress and adversity. The resilience scale is made up of 10 items, with a range of scores from 0 to 40, with higher scores indicating greater resilience.
  First measurement: Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 4 weeks after the first measurement the second measurement of the same variable was carried out.
  Third measurement: POST Up to 4 weeks after the second measurement the third measurement of the same variable was carried out.
Outcome Measure: Change in Perceived Importance of Health Habits (Baseline-Pre-Post) | Baseline up to 8 weeks
  A self-report questionnaire specifically developed for this study will be used to assess adolescents' perceived importance of maintaining healthy habits. The instrument consists of 16 Likert-type items (1 = Not important at all to 5 = Extremely important) that evaluate three domains:
  1. Nutrition (e.g., balanced diet, regular meal patterns).
  2. Hygiene (e.g., daily personal hygiene routines).
  3. Physical exercise (e.g., regular engagement in physical activity).
  4. Healthy sleep habits (e.g. sleeping at least 8 hours, having a defined schedule.) Higher scores indicate greater perceived importance attributed to healthy behaviors across the three domains, with a total score ranging from 16 to 80. Subscale scores will also be calculated for each domain.
  First measurement (T1): Baseline, after informed consent. Second measurement (T2): Approximately 4 weeks after baseline (pre-intervention re-assessment).
  Third measurement (T3): Approximately 4 weeks after T2 (post-intervention assessment)
Outcome Measure: Assessment of the intervention and change in the emotional state of the participants | Baseline up to 8 weeks
  These items aim to assess the intervention from the perspective of adolescents, specifically in terms of the extent to which it has helped them in different areas of their daily lives. There will be a total of 13 Likert-type items ranging from 0 (it has not helped me at all) to 10 (it has helped me a lot). These items will only be collected at the final time point (T3), i.e. after the intervention has been completed.
  The degree of difficulty experienced in their lives and their emotional state will also be evaluated using six Likert scale items ranging from 0 to 10. Information on these difficulties and emotional state assessments will be collected at the three assessment points (T1, T2 and T3).
  First measurement (T1): Baseline, after informed consent. Second measurement (T2): Approximately 4 weeks after baseline (pre-intervention re-assessment).
  Third measurement (T3): Approximately 4 weeks after T2 (post-intervention assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Marián Pérez-Marín, PHD, Principal Investigator — Universitat de Valencia
Locations (1):
- Facultat de Psicología, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No